CLINICAL TRIAL: NCT05441839
Title: UK Heart Failure With Preserved Ejection Fraction Registry
Brief Title: UK Heart Failure With Preserved Ejection Fraction
Acronym: UK HFpEF
Status: Recruiting | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Pumping Marvellous Foundation (Unknown); British Society for Heart Failure (Unknown); National Institute for Health Research, United Kingdom (Other Government); British Heart Foundation Data Science Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: B01434
Record Dates: First submitted 2022-05-26; First posted 2022-07-01 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFpEF)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling will be performed for DNA extraction, plasma and serum. The total volume of blood collected will be up to 50 ml. Samples will undergo initial processing and storage at sites, before being transferred to a central repository (NIHR National Biosample Centre). Further details regarding collection, initial processing and storage, and transfer of samples to the central repository will be provided in the Study Reference Manual.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure occurs when the heart is no longer able to pump blood around the body properly. It can cause breathlessness, swollen feet and ankles, and tiredness. In about half of patients with heart failure, one measure of the heart's pumping function, called the 'ejection fraction', is normal. This type of heart failure is called heart failure with preserved ejection fraction, or HFpEF.

HFpEF remains poorly understood. It is not clear why some people develop HFpEF, or what determines the severity of the condition. Treatment options may be limited.

UK HFpEF is a study that aims to gain a better understanding of why people develop HFpEF, develop better tests to diagnosis it, identify and test new treatments, and follow the health of the people taking part over many years.

DETAILED DESCRIPTION:
Approximately half of patients with heart failure have a normal, or preserved, left ventricular ejection fraction (HFpEF) (Owen et al, 2006). Rather than being a single diagnosis, it has become clear that HFpEF represents a heterogeneous syndrome involving a range of pathophysiological mechanisms, clinical factors and outcomes (Lewis et al, 2017). However, to-date, HFpEF has generally been considered as a single disease entity. Several high profile phase III trials in HFpEF have shown potentially impressive efficacy in some subgroups of patients, but failed to prove significance over entire cohorts (Pitt et al, 2014) (Solomon et al, 2019). This is likely due to the 'one-size-fits-all' approach taken, with insufficient stratification of the various underlying disease mechanisms.

The large and rapidly growing burden that HFpEF places on our healthcare systems mean there is a pressing need to better understand HFpEF and improve the management of patients with it. The recurrent lack of benefit of the one-size-fits-all approach mandates a new, personalised approach.

The UK HFpEF registry will be a key platform for collaborative UK clinical and translational HFpEF research. The aim is that multiple centres will collaborate and contribute patients such that the registry will provide deep phenotyping, linked to outcomes, in, ultimately, many thousands of patients. This will enable, for example, machine learning techniques to be applied at scale in order to reclassify HFpEF more powerfully. It will provide a platform for the development of diagnostics specific to the different HFpEF subgroups, and for more effective trials that will target groups of patients in whom new, repurposed or previously discarded treatments are expected to be effective. Moreover, it will provide cohorts of patients readily available for recruitment, with linkage in place for outcomes. It could be used to leverage commercial funding and participation, facilitated by simplified, single-point access for industry. It will enable scaled investigation aimed at understanding causes of HFpEF, improving risk stratification and providing better care.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Diagnosis of HFpEF by a cardiologist with HF expertise, or a primary care physician with HF expertise, or a heart failure nurse
3. Natriuretic peptide levels measured

Exclusion Criteria:

1. LV EF < 40% (at screening or any previous measurement)
2. Known infiltrative cardiomyopathy (e.g., amyloid, sarcoid, lymphoma, endomyocardial fibrosis)
3. Known active myocarditis, constrictive pericarditis, or cardiac tamponade
4. Known genetic hypertrophic cardiomyopathy or obstructive hypertrophic cardiomyopathy
5. Known arrhythmogenic right ventricular cardiomyopathy
6. Known severe primary valvular heart disease
7. Known idiopathic, heritable or drug-induced pulmonary arterial hypertension
8. Heart transplantation or ventricular assist device
9. Complex congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals will be considered for inclusion in this study regardless of age, disability, gender reassignment, marriage and civil partnership, pregnancy and maternity, race, religion and belief, sex, and sexual orientation, except where the study inclusion and exclusion criteria explicitly state otherwise.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2037-06-01 (Estimated); Study Completion 2037-06-01 (Estimated)

PRIMARY OUTCOMES:
Identification of distinct subgroups of HFpEF | 10 years
  Identify distinct subgroups of HFpEF based on disease mechanisms, clinical factors and outcomes
Improve understanding of the causes of HFpEF | 10 years
  Improve the understanding of the cause of HFpEF to provide the basis for developing and evaluating new therapies and diagnostics
Improve risk stratification of HFpEF | 10 years
  Identify and improve risk stratification models for HFpEF patients

CONTACTS AND LOCATIONS:
Overall Officials: Chris Miller, MBChB FRCP, Study Chair — Manchester University NHS Foundation Trust
Locations (26):
- United Kingdom (26):
  - Cwm Taf Morgannwg University Health Board, Abercynon
  - Buckinghamshire Healthcare NHS Trust, Aylesbury
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Broomfield Hospital, Chelmsford
  - NHS Tayside, Dundee
  - Glasgow Royal Infirmary, Glasgow
  - West Suffolk NHS Foundation Trust, Ipswich
  - Kettering General Hospital, Kettering
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Foundation Trust, Leicester
  - Barnet Hospital, London
  - Guys and St. Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Manchester University NHS Foundation trust, Manchester
  - The James Cook University Hospital, Middlesbrough
  - Northumbria Healthcare NHS Foundation Trust, Newcastle upon Tyne
  - Norfolk & Norwich University Hospitals NHS Foundation Trust, Norwich
  - George Eliot Hospital, Nuneaton
  - North West Anglia NHS Foundation Trust, Peterborough
  - University Hospitals Dorset NHS Foundation Trust, Poole
  - Betsi Cadwaldr University Health Board, Rhyl
  - Salisbury NHS Foundation Trust, Salisbury
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospital of North Tees, Stockton-on-Tees
  - South Tyneside & Sunderland NHS Foundation Trust, Sunderland
  - Southend University Hospital, Westcliff-on-Sea

IPD SHARING:
Plan to Share IPD: Yes
Participants will be asked to provide consent for pseudonymised study data, including, for example, individual patient-level data, scans and any other study data, to be shared for research purposes with investigators or organisations, including independent commercial organisations ('industry'), in the United Kingdom or overseas, including outside of the European Economic Area and in the United States of America. Participant personal details such as name, address, date of birth, will not be shared.
  Requests for access to the data will be managed by the Executive Steering Committee. Release of data to investigators or organisations requesting access, whether they reside within or outside the UK, will be covered by a Data Transfer Agreement. The Data Transfer Agreement is a legally binding document that will regulate the use of data to ensure that standards are maintained.
Time Frame: Within the life time of the study
Access Criteria: Release of data or samples to investigators or organisations requesting access, whether they reside within or outside the UK, will be covered by Data and/or Material Transfer Agreements. The Agreements are legally binding documents that will regulate the use of data and/or samples to ensure that standards are maintained.

REFERENCES:
- [Background] Owan TE, Hodge DO, Herges RM, Jacobsen SJ, Roger VL, Redfield MM. Trends in prevalence and outcome of heart failure with preserved ejection fraction. N Engl J Med. 2006 Jul 20;355(3):251-9. doi: 10.1056/NEJMoa052256. PMID 16855265
- [Background] Lewis GA, Schelbert EB, Williams SG, Cunnington C, Ahmed F, McDonagh TA, Miller CA. Biological Phenotypes of Heart Failure With Preserved Ejection Fraction. J Am Coll Cardiol. 2017 Oct 24;70(17):2186-2200. doi: 10.1016/j.jacc.2017.09.006. PMID 29050567
- [Background] Pitt B, Pfeffer MA, Assmann SF, Boineau R, Anand IS, Claggett B, Clausell N, Desai AS, Diaz R, Fleg JL, Gordeev I, Harty B, Heitner JF, Kenwood CT, Lewis EF, O'Meara E, Probstfield JL, Shaburishvili T, Shah SJ, Solomon SD, Sweitzer NK, Yang S, McKinlay SM; TOPCAT Investigators. Spironolactone for heart failure with preserved ejection fraction. N Engl J Med. 2014 Apr 10;370(15):1383-92. doi: 10.1056/NEJMoa1313731. PMID 24716680
- [Background] Solomon SD, McMurray JJV, Anand IS, Ge J, Lam CSP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Redfield MM, Rouleau JL, van Veldhuisen DJ, Zannad F, Zile MR, Desai AS, Claggett B, Jhund PS, Boytsov SA, Comin-Colet J, Cleland J, Dungen HD, Goncalvesova E, Katova T, Kerr Saraiva JF, Lelonek M, Merkely B, Senni M, Shah SJ, Zhou J, Rizkala AR, Gong J, Shi VC, Lefkowitz MP; PARAGON-HF Investigators and Committees. Angiotensin-Neprilysin Inhibition in Heart Failure with Preserved Ejection Fraction. N Engl J Med. 2019 Oct 24;381(17):1609-1620. doi: 10.1056/NEJMoa1908655. Epub 2019 Sep 1. PMID 31475794
- [Derived] UK HFpEF Collaborative Group. Rationale and design of the United Kingdom Heart Failure with Preserved Ejection Fraction Registry. Heart. 2024 Feb 12;110(5):359-365. doi: 10.1136/heartjnl-2023-323049. PMID 37827557